CLINICAL TRIAL: NCT06212024
Title: The Effectiveness of Mentalization-Based Treatment-Early (MBT-early) in Adolescents With Emerging Borderline-personality Disorder: a Single Case Experimental Design
Brief Title: MBT-early: a Single Case Experimental Design
Status: Active, not recruiting | Type: Observational
Sponsor: De Viersprong (Other)
Responsible Party: Sponsor
Other Study IDs: NL85140.028.23
Record Dates: First submitted 2023-12-13; First posted 2024-01-18 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline personality disorder; Early intervention; Single case experimental design; Treatment outcome
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MBT-early: See intervention description. Within subject comparison.
  Interventions: Behavioral: Mentalization Based Treatment-early

INTERVENTIONS:
Behavioral: Mentalization Based Treatment-early — MBT-early is an early intervention program for young people at risk for developing BPD that has been developed as an adaptation of MBT, an empirically supported treatment for BPD. MBT-early is a time-limited intervention that has been designed for early-stage BPD and focuses on improving personality functioning. MBT-early is a two-phase treatment that integrates interventions at the individual, family, and context level. MBT-early provides a combination of treatment modalities, including individual and family sessions, case management, and treatment reviews. Interventions are tailored to the specific needs of the young person and his/her family. The treatment consists of 16 weekly individual sessions, 3 family sessions, and case management. The initial treatment phase (16 weeks) is followed by a booster period (6 months) with 4 booster sessions. Since MBT-early involves a flexible approach, this standard package may be downscaled in cases of rapid improvement, or upscaled when needed.

SUMMARY:
Borderline personality disorder (BPD) is characterized by problems in emotion regulation, identity disturbances, and impaired interpersonal functioning. Because BPD may determine health and quality of life in long term, it is important to focus on early detection and early intervention to prevent worsening. In this study, the effectiveness of a new intervention, MBT-early, is investigated in adolescents with borderline personality problems, using a single-case experimental design (SCED).

V1.0 Initial release - [13/12/2023]: Initial registration.

V1.1 2 Amendments - [14-07-2025]:

* (1) Amendment to to clarify the use of diagnostic data (SCID-5-S) for inclusion purposes and to add logbooks documenting deviations from standard treatment protocols. Approved by the METC on 22-10-2024.
* (2) Amendment to include to expand the sample size from 6 to 8 participants and to include a qualitative component involving semi-structured interviews with participants, their caregivers, and therapists. Approved by the METC on 23-01-2025.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is characterized by problems in emotion regulation, identity disturbances, and impaired interpersonal functioning. Because BPD may determine health and quality of life in long term, it is important to focus on early detection and early intervention to prevent worsening. In this study, the effectiveness of a new intervention, MBT-early, is investigated in adolescents with borderline personality problems through a single case experimental design (SCED). Existing studies into the efficacy of psychotherapeutic interventions for young people with a (subclinical) borderline personality disorder (BPD) show mixed results. An obvious explanation therefore lies in the heterogeneity of the samples studied, where the same intervention is investigated by young people with some characteristics of borderline personality problems in an early stage as by young people with significant borderline personality problems at a later stage. However, there is evidence that interventions should be targeted specifically at the stage of progression of the disorder ('staged care'). Interventions may be more effective when they correspond to the stage of disease progression. MBT-early is an intervention intended for young people in an early stage of BPD. The intervention not only addresses the characteristics of BPD, but generally aims to improve personality functioning. MBT-early focuses on strengthening the young person's mentalizing capacity and to increase epistemic trust (the openness to learn from others) in order to prevent developmental stagnation and chronic consequences of personality disfunctioning. Although there is evidence for the efficacy of MBT for adults and adolescents, MBT-early has not yet been studied in terms of effectiveness. This study sets out to investigate the effectiveness of MBT-early, using a Single Case Experimental Design. The investigators hypothesize that treating youngsters with early features of BPD with MBT-early results in reduction of features of personality problems and the most frequently occurring symptoms (depressive symptoms). Exploratively mechanisms of change are being explored.

Research questions:

1. What is the effectiveness of MBT-early in youth with early stage BPD? 1a) What effect does MBT-early have on the improvement of personality functioning? 1b) What effect does early MBT have on the degree of depressed mood?
2. What are the possible working mechanisms of MBT-early? 2a) Does the youth's mentalizing ability influence the improvement of personality functioning? 2b) Does epistemic trust affect the improvement of personality functioning?

Objective of the study: The primary objective is to study the effectiveness of MBT-early in terms of treatment outcome on personality functioning and depressive symptoms. As a second objective the investigators will exploratively study the presumed working mechanisms of the MBT-early intervention (mentalizing capacities and epistemic trust).

Amendment 1 (Approved October 22, 2024):

Diagnostic information obtained during intake, using the Structured Clinical Interview for DSM-5 Syndrome Disorders (SCID-5-S), is used to verify inclusion criteria. Although this was part of the original protocol, it has now been explicitly clarified in the participant information material. Additionally, therapist-maintained logbooks documenting deviations from standard treatment protocols (e.g., missed sessions or clinical incidents) have been introduced to enhance contextual interpretation of the SCED data.

Amendment 2 (Approved January 23, 2025):

To increase the representativeness of the sample, the maximum number of participants has been increased from 6 to 8. Furthermore, a qualitative component was added to the design. After completing treatment, participants, their caregivers, and their therapists will be invited to take part in semi-structured interviews to explore perceived treatment processes and outcomes. These interviews aim to enrich interpretation of quantitative findings and explore perspectives on symptom change, treatment satisfaction, and contextual factors.

ELIGIBILITY:
Inclusion Criteria:

1. age between 12 and 18 years,
2. Three to six traits of borderline personality disorder as assessed by the Structured Clinical Interview for DSM-5 Syndrome Disorders
3. Mild to moderate disability with regard to functioning in school, at home and in the peer group.

Exclusion Criteria:

1. presence of a primary diagnosis that requires other specialist treatment (e.g. autism spectrum disorder, chronic psychotic disorder, severe eating disorder of sever substance abuse disorder),
2. More than one comorbid classification,
3. IQ < 75,
4. Severe disability with regard to functioning in school, at home and in the peer group representative for later stage BPD.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The target population of this study consists of adolescents referred to de Viersprong, with early-stage BPD, that are indicated for MBT-early by means of regular intake procedure. All adolescents referred to MBT-early are eligible for participation in the study, as there are no additional inclusion criteria for the study, aside from the clinical inclusions and exclusion criteria for the MBT-Early intervention
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Level of Personality Functioning | through study completion, approximately 1 year
  Assessed by the Level of Personality Functioning Scale-Brief form, version 2.0 (LPFS-BF-2.0, 12 items). Weekly assessment during the baseline period of six weeks, weekly assessment during the intervention period of 16 weeks and 4 assessments spread over a period of six months, during the booster phase.
Depressive symptoms | through study completion, approximately 1 year
  Assessed by the Patient Health Questionnaire-2 (PHQ-2, 2 items). Weekly assessment during the baseline period of six weeks, weekly assessment during the intervention period of 16 weeks and 4 assessments spread over a period of six months, during the booster phase.

SECONDARY OUTCOMES:
Mentalizing Capacities | through study completion, approximately 1 year
  Assessed by the Reflective Function Questionnaire for Youth-5 (RFQY-5). Weekly assessment during the baseline period of six weeks, weekly assessment during the intervention period of 16 weeks and 4 assessments spread over a period of six months, during the booster phase.
Epistemic Trust | through study completion, approximately 1 year
  Assessed by 4 selected items from the Questionnaire Epistemic Trust (QET). Weekly assessment during the baseline period of six weeks, weekly assessment during the intervention period of 16 weeks and 4 assessments spread over a period of six months, during the booster phase.

OTHER OUTCOMES:
Semi-structured interviews | Within 60 days after completion of Phase C (final intervention session)
  Qualitative data from semi-structured interviews with participants, caregivers, and therapists about perceived treatment effects, explanatory factors, and general experiences with MBT-early.
  Semi-structured qualitative interviews with adolescent participants, their caregivers, and their therapists will be conducted within a maximum of 60 days following the final intervention session (completion of Phase C). Interviews will be scheduled as soon as feasible after treatment completion, depending on participant availability, but will not exceed the 60-day time frame

CONTACTS AND LOCATIONS:
Overall Officials: Maaike L. Smits, PhD, Principal Investigator — Psychotherapeutisch centrum de Viersprong, te Halsteren
Locations (1):
- Psychotherapeutisch centrum de Viersprong, te Halsteren, Halsteren, Netherlands

IPD SHARING:
Plan to Share IPD: No